CLINICAL TRIAL: NCT00870753
Title: Yoga in Treatment of Eating Disorders
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Kari Ebbesen Karlsen, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2.2006.1243
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Eating Disorders
Keywords: Eating disorders; yoga; body awareness; depression; anxiety
MeSH Terms: conditions — Feeding and Eating Disorders; Depression; Anxiety Disorders | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental): 90 min hatha yoga 2 times per week for 12 weeks.
  Interventions: Behavioral: Yoga
- Controls (No Intervention): Control group are offered the yoga intervention after finishing the study

INTERVENTIONS:
Behavioral: Yoga — 90 min hatha yoga 2 times per week for 12 weeks.
  Arms: Yoga

SUMMARY:
Purpose: to examine effects of hatha yoga in treatment of eating disorders.

Methods:

Participants: patients with DSM-IV Anorexia Nervosa, Bulimia Nervosa or Eating Disorders Not Otherwise Specified will be invited to participate in this study. Exclusion criteria will be age under 18, serious medical complications, psychosis or increased risk of suicide.

Design: randomized controlled single-blinded trial. Intervention: 2 x 90 min weekly group sessions for 12 weeks with hatha yoga. Main outcome measure: reduction in Eating Disorders Examination score. Secondary outcome measures: reduction in body dissatisfaction, depression and anxiety

DETAILED DESCRIPTION:
For the last years, yoga has become a popular "body-mind" form of exercise in western countries (Daubenmier, 2005). Yoga has shown good effects on increasing muscle strength, flexibility and stability, in addition studies have found reduced stress level, improved mood and breathing (Astin et al., 2003; Gimbel, 1998b; Granath et al., 2006; Lavey et al., 2005; Manjunatha et al., 2005b; Netz & Lidor, 2003a; Telles & Naveen, 1997b; Yadav et al., 2005b). Previous research have shown a tendency for persons practicing yoga improving body awareness and body sensitivity, and reduction of body dissatisfaction (Daubenmier, 2005). In addition, two studies have examined yoga in treatment of binge eating disorder (Daubenmier, 2005; Gimbel, 1998a). Results showed reduction in number of binge eating episodes in the intervention group compared to the control group. No available studies have examined effect of yoga in treatment of the eating disorders types Anorexia Nervosa or Bulimia Nervosa.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or above
* DSM-IV Anorexia nervosa, Bulimia nervosa or Eating disorders not otherwise specified

Exclusion Criteria:

* serious medical complications
* psychosis
* suicidal behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
reduction in eating disorders symptoms assessed by Eating Disorders Examination clinical interview | after 12 weeks

SECONDARY OUTCOMES:
increased body awareness | after 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Oslo County, Norway